CLINICAL TRIAL: NCT03751722
Title: Genetic an Functional Studies of Patient With Inflammatory Bowel Disease
Acronym: MINOTOR
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2005/0528; DGS 2006/0083 (Other: Number reference,Ministry of health)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn disease; Ulcerative colitis; genetic makers; cytokines
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to study the response of macrophages, isolated from patients with ulcerative colitis (Crohn's disease) or Crohn's disease (CD), to 6 candidate enterogenous and their derivatives, depending on the genotype for associated polymorphisms. to the development of IBD

ELIGIBILITY:
Inclusion Criteria:

* patient with definite crohn's disease or ulcerative colitis

Exclusion Criteria:

* patient receiving anti-TNF therapy during 14 days before inclusion.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All outpatients and inpatients from gastroenterology units of adulte and pediatric references centers
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Isolated macrophage response measured by PCR | Baseline: one session
  identification of macrophage activation markers specific analysis of gene expression (by PCR in real time) and / or the production (ELISA) of proinflammatory molecules (IL-6, TNF-1 and IL-8), anti-inflammatory (IL-10) and immunomodulatory (IL4,PPAR -2, MOR)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Gower-Rousseau, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No